CLINICAL TRIAL: NCT02450071
Title: Pre-Hospital Advanced Airway Management in the Nordic Countries - A Prospective Multicentre Observational Study
Brief Title: Pre-Hospital Advanced Airway Management in the Nordic Countries
Acronym: PHAST
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Principal Investigator, Mikael Gellerfors, MD, Karolinska Institutet
Other Study IDs: PHAST-01
Record Dates: First submitted 2015-05-07; First posted 2015-05-21 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest; Trauma; Traumatic Brain Injury; Hypoventilation; Airway Obstruction; Emergencies
Keywords: Pre-hospital; Out-of-hospital; Prehospital emergency care (MeSH); Emergency medical services (MeSH); Helicopter emergency medical service; Critical care (MeSH); Airway management (MeSH); Endotracheal intubation (MeSH); Difficult endotracheal intubation; Complications (MeSH); Patient safety
MeSH Terms: conditions — Heart Arrest; Wounds and Injuries; Brain Injuries, Traumatic; Hypoventilation; Airway Obstruction; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pre-Hospital Advanced Airway Management (PHAAM) is a potentially lifesaving intervention. A recent Danish multicentre single country study demonstrated a 99,7% incidence of successful anaesthesiologist pre-hospital endotracheal intubation, with a PHAAM-related complication rate of 7.9%. A London study revealed a significantly higher intubation failure rate among non-anaesthesiologist physicians. In Scandinavia different types of emergency medical services (EMS) and professions provide PHAAM. The success rate of prehospital endotracheal intubation (PHETI), incidence of difficult intubation and complications in the Nordic countries is not known. The aim of this study is to define PHAAM success rate and complications in different types of Nordic EMS organisations and physician critical care teams. The study is a prospective observational study with collection of PHAAM data according to the template by Sollid et al. in the 12 participating Nordic Countries EMS/HEMS centres and physician critical care teams. The primary endpoint is PHETI success on ≤2 attempts and no complications.

DETAILED DESCRIPTION:
Pre-Hospital Advanced Airway Management (PHAAM) is a potentially lifesaving intervention. A recent meta-analysis of >15.000 patients reported a variation in the prehospital endotracheal intubation (PHETI) success rate with different methods used and provider background. A recent prehospital study from London revealed a significantly higher intubation failure rate among non-anaesthesiologist physicians. In Scandinavia different types of emergency medical services (EMS) and professionals provide PHAAM. The success rate of PHETI, incidence of difficult intubation and complications in the Nordic countries is not known. Although the EMS structure in Scandinavia is reasonably similar, there are some inter- and intra-national differences regarding mission profile, staffing, systems for dispatch and on-scene management. A Danish PHAAM study demonstrated a 99,7% anaesthesiologist PHETI success rate with a 7,9% complication rate. The authors concluded the study was from a homogenous Danish system limiting the ability to generalise the findings to other systems with different staffing, caseload or case mix.

The PHAST investigators aim to provide prospective multicentre data on the pre-hospital intubation success rate and complications in the Nordic countries. Additionally the investigators will compare the PHAAM procedure for different subgroups of patients, regions and EMS organisations.

In the PHAST observational study twelve Nordic (Sweden, Norway, Denmark and Finland) Helicopter and Rapid Response Emergency Medical Services will include patients during 18 months. The decision to perform PHAAM is based on the discretion of prehospital provider. The PHAAM core data will be prospectively collected according the template by Sollid et al.

The primary endpoint is PHETI success on ≤2 attempts and no complications. Secondary endpoints include overall PHETI success rate, PHETI success on 1st, 2nd, 3rd and >3rd attempt, difficult PHETI, success rate of laryngeal mask and surgical airway, PHAAM complications and prehospital mortality.

Through predefined analysis of the data, the PHAST investigators hope to

1. Describe the characteristics and outcome of advanced prehospital airway management.
2. Identify which groups of critically injured or ill patients will benefit most from competent advanced prehospital airway management, and identify specific areas for future research.

ELIGIBILITY:
Inclusion Criteria:

All patients requiring prehospital advanced airway management (PHAAM) by the Helicopter Emergency Medical Services (EMS) and Ground EMS (GEMS) units in the study. PHAAM includes endotracheal intubation, supraglottic airway and percutaneous/surgical airway. The indications for performing PHAAM as categorised by Sollid et al. are

* Decreased level of consciousness
* Hypoxemia
* Ineffective ventilation
* Existing airway obstruction
* Impending airway obstruction
* Combative or uncooperative patient
* Relief of pain or distress
* Cardiopulmonary arrest
* Other

Exclusion Criteria:

* Patients receiving advanced airway management during so-called secondary missions (or inter-hospital transfer)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients requiring prehospital advanced airway management (PHAAM) by the Helicopter Emergency Medical Services (EMS) and Ground EMS (GEMS) units in the study. PHAAM includes endotracheal intubation, supraglottic airway and percutaneous/surgical airway.
Sampling Method: Probability Sample
Enrollment: 2028 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
PHETI ≤ 2attempts and no complications | At hospital admission (</= 1 day)
  Prehospital Endotracheal Intubation success and complications as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)

SECONDARY OUTCOMES:
PHETI overall success rate | At hospital admission (</= 1 day)
  PHETI= Prehospital Endotracheal Intubation as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
PHETI success on 1st attempt and no complications | At hospital admission (</= 1 day)
  Endpoint as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
PHETI success rate on 1st, 2nd, 3rd and >3rd attempt | At hospital admission (</= 1 day)
  PHETI success as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
PHAAM Complications | At hospital admission (</= 1 day)
  PHAAM Complications as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
Success rate of airway back-up devices | At hospital admission (</= 1 day)
  Endpoint as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
Pre-hospital mortality | At hospital admission (</= 1 day)
  Endpoint as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
Other pre-specified endpoints and analysis as defined by the ERB-submitted protocol | At hospital admission (</= 1 day)
  Endpoints as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)
Mortality | At hospital discharge (estimated average 7 days)
Mortality | At 30 days
PHETI ≤ 2attempts and no complications among patients with TBI | At hospital discharge (estimated average 7 days)
  PHETI ≤ 2attempts and no complications among subgroup of patients with Traumatic Brain Injury. Prehospital Advanced Airway Management (PHAAM) success and complications as defined by Sollid et al (Sollid SJ, Lockey D, Lossius HM: A consensus-based template for uniform reporting of data from pre-hospital advanced airway management. Scand J Trauma Resusc Emerg Med 2009, 17:58.)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Morten Lossius, MD, PhD, Study Chair — Norwegian Air Ambulance Foundation
Locations (1):
- HEMS VGR, Gothenburg, VästraGötaland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided